CLINICAL TRIAL: NCT06114160
Title: Knowledge of Pregnant Women Concerning Pertussis, Vaccination Against Pertussis and Cocooning Strategy
Acronym: Coqueluche-Vac
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_015_Coqueluche-Vac
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Pertussis
Keywords: cocooning strategy; pertussis; pregnancy; vaccination against pertussis
MeSH Terms: conditions — Whooping Cough | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women: Pregnant women between 20 and 41 weeks of amenorrhoea, primiparous.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
In France, it has been recommended since 2022 that pregnant women be vaccinated against pertussis from 20 to 36 weeks' gestation.

This vaccination schedule is inspired by the Anglo-Saxon model and studies showing the effectiveness of this practice.

The aim of this vaccine is to protect the newborn by transferring antibodies from the fetus to the placenta, because Pertussis is a particularly serious disease in newborns.

DETAILED DESCRIPTION:
The aim is to describe pregnant women's knowledge concerning pertussis, vaccination against pertussis during pregnancy and the cocooning strategy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant between 20 and 41 weeks of amenorrhea
* Primiparous
* aged more than 18
* Agreed to participate in the study

Exclusion Criteria:

* Multiparous
* Protected by law (guardianship, guardianship, safeguarding of justice)
* Not agreed to participate in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
recommendation of vaccination against pertussis | day0
  Knowledge of pregnant women's concerning recommendation of vaccination against pertussis from 20 to 36 weeks' gestation : does the woman know or not the recommandation concerning the vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pilet Caroline, midwife, Principal Investigator — CHU de Reims

IPD SHARING:
Plan to Share IPD: Undecided